CLINICAL TRIAL: NCT01814293
Title: Comparison of Supportive Therapies for Symptom Relief From Pediatric Upper Respiratory Infections (URIs)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: loss of funding. No data was collected.
Sponsor: University of California, San Francisco (Other)
Collaborators: Vapore, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 12-10271
Record Dates: First submitted 2013-03-13; First posted 2013-03-19 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Acute Upper Respiratory Infection; Signs and Symptoms
Keywords: Pediatric; Upper Respiratory infection; Over the Counter Drugs; Drugs, Non-Prescription; Vaporizer
MeSH Terms: conditions — Signs and Symptoms; Respiratory Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Handheld humidifier (Active Comparator): Study design is a nonblinded randomized controlled comparison study of pediatric patients presenting to the UCSF Emergency Department (ED) with upper respiratory infection (URI) symptoms for which the ED physician has recommended supportive care only (ie. non-prescription symptom relief). Subjects will be randomized into 2 groups: handheld humidifier group (FDA cleared medical device that uses distilled water) & control group. Both groups may use any supportive modalities desired such as over-the-counter cold medications (OTCs), room air humidifier etc. Follow up surveys will be obtained on days 1 and 2 following the ED visit to assess whether then intervention (use of handheld humidifier) improved symptom scores or reduced the use of OTC medications or room humidifier.
  Interventions: Device: Handheld humidifier
- Control group (No Intervention): Subjects will manage cold symptoms with any desired supportive over the counter treatment, and complete surveys related to symptom scores and modalities used.

INTERVENTIONS:
Device: Handheld humidifier — Subjects will be randomized into 2 groups: handheld humidifier group (FDA cleared medical device that uses distilled water) & control group. Both groups may use any supportive modalities desired such as over-the-counter cold medications (OTCs), room air humidifier etc. Follow up surveys will be obtained on days 1 and 2 following the ED visit to assess whether then intervention (use of handheld humidifier) improved symptom scores or reduced the use of OTC medications or room humidifier.
  Other Names: MyPurMist (specific handheld humidifier used in this trial)
  Arms: Handheld humidifier

SUMMARY:
This is a nonblinded randomized controlled trial which is a survey-based comparison between supportive treatments for symptom relief from pediatric upper respiratory infection (URI). The primary objective of this study is to determine if the use of handheld humidifier improves URI symptom scores and/or reduces use of over the counter medications compared to other supportive treatments for pediatric URIs (ie. OTC cold medications, room air humidifier). Study duration is approximately 1 year and the individual intervention is 4 days.

DETAILED DESCRIPTION:
Study design is a nonblinded randomized controlled trial. It is a survey-based comparison study of pediatric patients presenting to the Emergency Department (ED) with upper respiratory infection (URI) symptoms for which the ED physician has recommended supportive care only (ie. non-prescription symptom relief). Study duration is approximately one year. Subject participation duration is 4 days.

Subjects will be randomized into 2 groups: handheld humidifier group (FDA cleared medical device that uses distilled water) & control group. Both groups may use any supportive modalities desired such as over-the-counter cold medications (OTCs), room air humidifier etc.

Primary study objective is to determine if the use of handheld humidifier improves URI symptom scores (nocturnal cough, parental perception) and/or reduces use of other supportive modalities compared to the control group for the relief of pediatric URI symptoms.

Three surveys will be obtained from all subjects. The initial survey occurs at the time of enrollment (T0). The second and third surveys will be completed by the parent/guardian on line or by phone on the first day after ED visit (T-1) and sometime between the 2nd-4th day after ED visit (T-2). The survey component includes a validated pediatric cough questionnaire with 7 point Likert scale, and a questions regarding any other supportive treatments used for symptom relief (the type, frequency and results).

ELIGIBILITY:
Inclusion Criteria:

* Ages 0-18 years old
* URI symptoms of less than 1 week duration.
* No new medications prescribed during this ED visit other than antipyretics and refills of routine medications (ie. refills of bronchodilators are OK).
* Symptom severity scores of atleast 3 ("sometimes" on a Likert 7 point scale) on at least 2 survey questions related to symptom scores (cough frequency/severity, effect on the child's sleep, effect on parental sleep, combined symptom severity).
* Parent consenting the child must have two valid forms of contact information (ie. phone number and email address) in order to follow up as needed for completion of 2nd and 3rd surveys.
* Parent consenting the child must have access to internet connection or phone for the following 2-4 days after enrollment.
* Parent consenting the child must be able to fluently read and speak English without the use of aides. This study budget does not allow for multilingual resources.

Exclusion Criteria:

* Chronic pulmonary disease
* Chronic or congenital cardiac disease
* Chronic cough
* Acute pneumonia
* Any patient that will receive a new prescription from this ED visit (antibiotics, inhalers, steroids, etc)
* Any patient currently using a handheld humidifier for this URI.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
URI (upper respiratory infection) symptoms one day after ED visit | 1 day
  Differences in symptom scores will be compared between handheld humidifier group and control group based on supportive treatments used. Proposed outcome is that the humidifier group has improved symptom scores and/or reduced use of other supportive modalities (ie. cold meds) compared to the control group during the time frame between the ED visit to the following day.
URI (upper respiratory infection) symptoms 2 days after ED visit | 1 day
  Differences in symptom scores will be compared between handheld humidifier group and control group based on supportive treatments used. Proposed outcome is that the humidifier group has improved symptom scores and/or reduced use of other supportive modalities (ie. cold meds) compared to the control group during the time frame between the 1st and 2nd days following the ED visit.

SECONDARY OUTCOMES:
URI (upper respiratory infection) revisits | 2 days
  Comparison between handheld humidifier group and control group regarding each group's symptom scores and need for revisits for same URI. Potential additional findings may include reduction of revisits for same URI, parental observed reduction in severity and/or duration of illness.

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline A Nemer, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Gunn VL, Taha SH, Liebelt EL, Serwint JR. Toxicity of over-the-counter cough and cold medications. Pediatrics. 2001 Sep;108(3):E52. doi: 10.1542/peds.108.3.e52. PMID 11533370
- [Background] Kuehn BM. FDA: cold medications risky for young children. JAMA. 2007 Sep 12;298(10):1151. doi: 10.1001/jama.298.10.1151. No abstract available. PMID 17848645
- [Background] Vernacchio L, Kelly JP, Kaufman DW, Mitchell AA. Pseudoephedrine use among US children, 1999-2006: results from the Slone survey. Pediatrics. 2008 Dec;122(6):1299-304. doi: 10.1542/peds.2008-0284. PMID 19047249
- [Background] Lokker N, Sanders L, Perrin EM, Kumar D, Finkle J, Franco V, Choi L, Johnston PE, Rothman RL. Parental misinterpretations of over-the-counter pediatric cough and cold medication labels. Pediatrics. 2009 Jun;123(6):1464-71. doi: 10.1542/peds.2008-0854. PMID 19482755
- [Background] Paul IM, Yoder KE, Crowell KR, Shaffer ML, McMillan HS, Carlson LC, Dilworth DA, Berlin CM Jr. Effect of dextromethorphan, diphenhydramine, and placebo on nocturnal cough and sleep quality for coughing children and their parents. Pediatrics. 2004 Jul;114(1):e85-90. doi: 10.1542/peds.114.1.e85. PMID 15231978
- [Background] Centers for Disease Control and Prevention (CDC). Infant deaths associated with cough and cold medications--two states, 2005. MMWR Morb Mortal Wkly Rep. 2007 Jan 12;56(1):1-4. PMID 17218934
- [Background] Dart RC, Paul IM, Bond GR, Winston DC, Manoguerra AS, Palmer RB, Kauffman RE, Banner W, Green JL, Rumack BH. Pediatric fatalities associated with over the counter (nonprescription) cough and cold medications. Ann Emerg Med. 2009 Apr;53(4):411-7. doi: 10.1016/j.annemergmed.2008.09.015. Epub 2008 Dec 19. PMID 19101060
- [Background] Rimsza ME, Newberry S. Unexpected infant deaths associated with use of cough and cold medications. Pediatrics. 2008 Aug;122(2):e318-22. doi: 10.1542/peds.2007-3813. PMID 18676517
- [Background] Daftary AS, Deterding RR. Inhalational lung injury associated with humidifier "white dust". Pediatrics. 2011 Feb;127(2):e509-12. doi: 10.1542/peds.2010-1312. Epub 2011 Jan 3. PMID 21199854
- [Background] Muller-Wening D, Koschel D, Stark W, Sennekamp HJ. [Humidifier-associated disease in the general population]. Dtsch Med Wochenschr. 2006 Mar 10;131(10):491-6. doi: 10.1055/s-2006-932548. German. PMID 16511738
- [Background] Baur X, Behr J, Dewair M, Ehret W, Fruhmann G, Vogelmeier C, Weiss W, Zinkernagel V. Humidifier lung and humidifier fever. Lung. 1988;166(2):113-24. doi: 10.1007/BF02714035. PMID 3130530
- [Background] Wallis BA, Turner J, Pearn J, Kimble RM. Scalds as a result of vapour inhalation therapy in children. Burns. 2008 Jun;34(4):560-4. doi: 10.1016/j.burns.2007.07.016. Epub 2007 Oct 22. PMID 17954012
- [Background] Donnelly D, Everard MM, Chang AB. Indoor air modification interventions for prolonged non-specific cough in children. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD005075. doi: 10.1002/14651858.CD005075.pub2. PMID 16856075